CLINICAL TRIAL: NCT00004259
Title: A Phase III Randomized Study (Phase I Closed) of Radiation Therapy and Temozolomide Versus Radiation Therapy and Nitrosourea for Anaplastic Astrocytoma And Mixed Anaplastic Oligoastrocytoma (Astrocytoma Dominant)
Brief Title: Radiation Therapy Combined With Chemotherapy in Treating Patients With Anaplastic Astrocytoma or Mixed Gliomas
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); North Central Cancer Treatment Group (Network); Eastern Cooperative Oncology Group (Network); NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RTOG-9813; CDR0000067512; ECOG-R9813; NCCTG-RTOG-9813
Record Dates: First submitted 2000-01-28; First posted 2003-01-27 (Estimated); Results first posted 2017-11-13 (Actual); Last update posted 2019-09-12 (Actual); Status verified 2019-08

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult anaplastic astrocytoma; adult mixed glioma
MeSH Terms: conditions — Central Nervous System Neoplasms; Astrocytoma; Glioma | interventions — Carmustine; Temozolomide; Radiotherapy; Lomustine

STUDY DESIGN:
Intervention Model Description: Phase I (sequential) followed by phase III (parallel)
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Radiation therapy + temozolomide (TMZ) (Experimental): Radiation therapy (RT) for 6 weeks concurrent with and followed by TMZ 200mg/m2 for twelve 28-day cycles
  Interventions: Drug: TMZ 200mg/m2; Radiation: radiation therapy
- RT + BCNU/CCNU (Active Comparator): Radiation therapy for 6 weeks concurrent with and followed by BCNU 80mg/m2 or CCNU 130 mg/m2 for six 8-week cycles
  Interventions: Drug: BCNU 80mg/m2; Radiation: radiation therapy; Drug: CCNU
- Pilot Arm #1: RT+TMZ+BCNU (Experimental): Radiation therapy for 6 weeks concurrent with and followed by BCNU 200mg/m2 and TMZ 150mg/m2 six 6-week cycles
  Interventions: Radiation: radiation therapy; Drug: BCNU 200mg/m2; Drug: TMZ 150mg/m2 six 6-week cycles
- Pilot Arm #2: RT+TMZ+BCNU (Experimental): Radiation therapy for 6 weeks concurrent with and followed by BCNU 150mg/m2 and TMZ 150mg/m2 six 8-week cycles
  Interventions: Radiation: radiation therapy; Drug: BCNU 150mg/m2; Drug: TMZ 150mg/m2 six 8-week cycles

INTERVENTIONS:
Drug: BCNU 80mg/m2 — BCNU 80 mg/m2 will be administered as an intravenous infusion on days 1, 2, and 3 of the first week of radiotherapy and on days 56, 57, and 58, then every eight weeks for four more cycles for a total of 6 cycles (maximum BCNU dose 1440 mg/m2).
  Arms: RT + BCNU/CCNU
Drug: TMZ 200mg/m2 — 200 mg/m2 orally on days 1-5 of the first week of radiotherapy. Repeat every 28 days for a total of 12 cycles.
  Arms: Radiation therapy + temozolomide (TMZ)
Radiation: radiation therapy — 1.8 Gy fractions (to isocenter), 1 fraction per day, 5 days per week to a dose of 59.4 Gy in 33 fractions.
Drug: CCNU — CCNU at 130 mg/m2 orally every 8 weeks for a total of 6 cycles. Administered on day 1 of the first week of radiotherapy and on day 56, then administered every 8 weeks for four more cycles for a total of 6 cycles.
  Arms: RT + BCNU/CCNU
Drug: BCNU 150mg/m2 — BCNU 150 mg/m2 will be administered as an intravenous infusion on day 5 of radiotherapy, and it will be repeated every eight weeks for a total of six cycles (maximum total BCNU dose 900 mg/m2).
  Arms: Pilot Arm #2: RT+TMZ+BCNU
Drug: BCNU 200mg/m2 — BCNU 200 mg/m2 will be administered as an intravenous infusion on day 1 of radiotherapy and will be repeated every six weeks for a total of 6 cycles (maximum BCNU dose 1200 mg/m2).
  Arms: Pilot Arm #1: RT+TMZ+BCNU
Drug: TMZ 150mg/m2 six 6-week cycles — 150 mg/m2 orally on days 1-5 of the first week of radiotherapy. Repeat for a total of six 6-week cycles
  Arms: Pilot Arm #1: RT+TMZ+BCNU
Drug: TMZ 150mg/m2 six 8-week cycles — 150 mg/m2 orally on days 1-5 of the first week of radiotherapy. Repeat for a total of six 8-week cycles
  Arms: Pilot Arm #2: RT+TMZ+BCNU

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Drugs used in chemotherapy, such as temozolomide, carmustine, and lomustine, use different ways to stop tumor cells from dividing so they stop growing or die. Combining radiation therapy with chemotherapy may kill more tumor cells.

PURPOSE: This randomized phase III trial is studying radiation therapy and temozolomide to see how well they work compared to radiation therapy and carmustine or lomustine in treating patients with anaplastic astrocytoma or mixed gliomas.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the overall survival and time to tumor progression in patients with anaplastic astrocytoma or mixed gliomas treated with radiotherapy combined with temozolomide vs carmustine or lomustine vs temozolomide and carmustine (arm discontinued as of 8/15/02).
* Compare the relative toxic effects of these regimens in these patients.
* Correlate molecular analyses with overall survival and time to tumor progression in patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to age (under 50 vs 50 and over), Karnofsky performance status (60-80% vs 90-100%), and prior surgery (biopsy only vs resection).

Phase I

* Pilot Arms I and II: Prior to initiating the randomization to 1 of 3 treatment arms in phase III, Patients are accrued to Arm III regimen to determine tolerability.

Phase III

* Patients are randomized to 1 of 2 treatment arms (3rd arm was dropped).

  * Arm I: Patients undergo radiotherapy 5 days a week for 6 weeks. Patients receive oral temozolomide on days 1-5 of the first week of radiotherapy. Chemotherapy repeats every 4 weeks for a total of 12 courses.
  * Arm II: Patients undergo radiotherapy as in arm I. Patients receive carmustine IV or lomustine IV over 1-2 hours on days 1-3 of the first week of radiotherapy and a second course on days 56-58. Chemotherapy repeats every 8 weeks for a total of 6 courses.
  * Arm III (dropped, did not open): Patients undergo radiotherapy as in arm I. Patients receive carmustine IV or lomustine IV over 3 hours on day 5 and oral temozolomide (2 hours after completion of carmustine or lomustine infusion) on days 1-5 of the first week of radiotherapy. Combination chemotherapy repeats every 8 weeks for 6 courses.

Patients are followed every 3 months for 1 year, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: Phase I: 30 patients; Phase III: 454 patients (227 per treatment arm) within 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven unifocal anaplastic astrocytoma or mixed gliomas, including the following:

  * Anaplastic astrocytoma
  * Mixed oligodendroglial/astrocytic tumors

    * Oligodendroglial component must be no greater than 25%
* No vascular proliferation and necrosis
* Increased cellularity, pleomorphism, and nuclear atypia allowed
* No tumor predominantly located in the posterior fossa (i.e., brainstem or cerebellum)
* Patients with prior biopsy proven low grade astrocytoma who now have anaplastic astrocytoma and have had no prior radiotherapy or chemotherapy also eligible
* Study therapy must begin within 6 weeks of diagnosis
* No spinal cord tumors, spinal drop metastases, or metastases to noncontiguous meninges

  * Pathologic evidence of local meningeal infiltration by underlying tumor allowed

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* At least 1 year

Hematopoietic:

* Hemoglobin at least 10 g/dL
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 150,000/mm^3

Hepatic:

* Bilirubin less than 2 times upper limit of normal (ULN)
* Aspartate aminotransferase (AST) less than 2 times ULN
* Alkaline phosphatase less than 2 times ULN

Renal:

* Blood urea nitrogen no greater than 25 mg/dL
* Creatinine less than 1.5 times normal

Pulmonary:

* No pre-existing lung disease that, in the investigator's opinion, would preclude administration of carmustine or lomustine or completion of therapy

Other:

* No other major medical illness or psychiatric impairment that would preclude study compliance
* No other malignancy within the past 5 years except nonmelanomatous skin cancer or carcinoma in situ of the cervix
* No known hypersensitivity to 1 of the components of carmustine, lomustine, temozolomide, dacarbazine, or any other nitrosourea
* No active infection
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior biologic therapy

Chemotherapy:

* See Disease Characteristics
* No prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics
* No prior radiotherapy to brain or head and neck

Surgery:

* Not specified

Other:

* No other concurrent anticancer treatment for anaplastic astrocytoma until a recurrence is detected

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2000-06; Primary Completion 2015-02-01 (Actual); Study Completion 2018-05-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan M. Chang, MD, Study Chair — University of California, San Francisco; Kurt A. Jaeckle, MD, Study Chair — Mayo Clinic; Peter Bushunow, MD, Study Chair — Lipson Cancer and Blood Center at Rochester General Hospital
Locations (92):
- United States (92):
  - Mobile Infirmary Medical Center, Mobile, Alabama
  - Arizona Oncology Services Foundation, Phoenix, Arizona
  - Enloe Cancer Center at Enloe Medical Center, Chico, California
  - North Bay Cancer Center, Fairfield, California
  - Solano Radiation Oncology Center, Vacaville, California
  - Lynn Regional Cancer Center at Boca Raton Community Hospital - Main Center, Boca Raton, Florida
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - Baptist Cancer Institute - Jacksonville, Jacksonville, Florida
  - Florida Oncology Associates at Southside Cancer Center, Jacksonville, Florida
  - Baptist Medical Center South, Jacksonville, Florida
  - Integrated Community Oncology Network, Jacksonville Beach, Florida
  - Florida Oncology Associates, Orange Park, Florida
  - Florida Cancer Center - Palatka, Palatka, Florida
  - Flagler Cancer Center, Saint Augustine, Florida
  - H. Lee Moffitt Cancer Center and Research Institute at University of South Florida, Tampa, Florida
  - John B. Amos Cancer Center, Columbus, Georgia
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Galesburg Clinic, Galesburg, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - InterCommunity Cancer Center of Western Illinois, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hopedale Medical Complex, Hopedale, Illinois
  - Kewanee Hospital, Kewanee, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - St. Margaret's Hospital, Spring Valley, Illinois
  - Valley Cancer Center, Spring Valley, Illinois
  - McFarland Clinic, PC, Ames, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cotton-O'Neil Cancer Center, Topeka, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - St. John's Regional Health Center, Springfield, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Deaconess Billings Clinic - Downtown, Billings, Montana
  - Good Samaritan Cancer Center at Good Samaritan Hospital, Kearney, Nebraska
  - Methodist Cancer Center at Methodist Hospital - Omaha, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Fox Chase Virtua Health Cancer Program at Virtua Memorial Hospital Marlton, Marlton, New Jersey
  - Franklin & Edith Scarpa Regional Cancer Center at South Jersey Healthcare, Vineland, New Jersey
  - Fox Chase Virtua Health Cancer Program at Virtua West Jersey, Voorhees Township, New Jersey
  - Lipson Cancer and Blood Center at Rochester General Hospital, Rochester, New York
  - Mission Hospitals - Memorial Campus, Asheville, North Carolina
  - Akron City Hospital, Akron, Ohio
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Case Comprehensive Cancer Center, Cleveland, Ohio
  - Cancer Research UK Medical Oncology Unit at Churchill Hospital & Weatherall Institute of Molecular Medicine - Oxford, Salem, Ohio
  - Cancer Treatment Center, Wooster, Ohio
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Allegheny Cancer Center at Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Reading Hospital and Medical Center, Reading, Pennsylvania
  - Guthrie Cancer Center at Guthrie Clinic Sayre, Sayre, Pennsylvania
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Latter Day Saints Hospital, Salt Lake City, Utah
  - Theda Care Cancer Institute, Appleton, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Community Memorial Hospital Cancer Care Center, Menomonee Falls, Wisconsin
  - University of Wisconcin Cancer Center at Aspirus Wausau Hospital, Wausau, Wisconsin

REFERENCES:
- [Result] Chang SM, Seiferheld W, Curran W, Share R, Atkins J, Choucair A, Kresl J, Thoron L, Cairncross G, Gilbert M, Bahary JP, Dolinskas C, Louis DN, Bushunow P, Buckner J, Barger G, Mehta M. Phase I study pilot arms of radiotherapy and carmustine with temozolomide for anaplastic astrocytoma (Radiation Therapy Oncology Group 9813): implications for studies testing initial treatment of brain tumors. Int J Radiat Oncol Biol Phys. 2004 Jul 15;59(4):1122-6. doi: 10.1016/j.ijrobp.2004.01.002. PMID 15234047

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Radiation Therapy + Temozolomide (TMZ) | RT + BCNU/CCNU | Pilot Arm #1: RT+TMZ+BCNU | Pilot Arm #2: RT+TMZ+BCNU
Started | 98 | 103 | 15 | 14
Completed | 97 | 99 | 15 | 14
Not Completed | 1 | 4 | 0 | 0
Not completed — Protocol Violation | 1 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Eligible patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Radiation Therapy + Temozolomide (TMZ) | RT + BCNU/CCNU | Pilot Arm #1: RT+TMZ+BCNU | Pilot Arm #2: RT+TMZ+BCNU | Total
Number analyzed (Participants) | 97 | 99 | 15 | 14 | 225
Age, Continuous [Median (Full Range); unit: years] | 42 [18 to 73] | 43 [19 to 80] | 48 [26 to 80] | 41 [25 to 74] | 43 [18 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 47 | 5 | 6 | 100
  Male | 55 | 52 | 10 | 8 | 125

OUTCOME MEASURES:

1. Primary Outcome: (Phase III) Overall Survival (OS)
Description: Survival time is defined as time from randomization to date of death from any cause and is estimated by the Kaplan-Meier method. Patients last known to be alive are censored at the date of last contact. Per the protocol, the pilot arms were not included in the Phase III analyses.
Time Frame: From randomization to date of death. Patients are followed until death. Analysis occurs after 155 deaths have been reported, estimated at 5.5 years from the study opening.
Population: Eligible randomized patients
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Radiation Therapy + Temozolomide (TMZ) | RT + BCNU/CCNU
Number analyzed (Participants) | 97 | 99
years | 3.9 [3.0 to 7.0] | 3.8 [2.2 to 7.0]
Statistical Analysis 1: Comparison: Radiation Therapy + Temozolomide (TMZ) vs RT + BCNU/CCNU; The hypothesized median survival time was 36 months for the RT+BCNU/CCNU arm and 54 months for the RT+TMZ arm, corresponding to a hazard ratio (HR) of 0.67. A sample size of 216 evaluable patients per arm would provide 90% power with a one-sided significance level of 0.05. The final analysis was planned after 155 deaths were observed. Interim efficacy analyses were planned after 52 and 104 deaths, with an interim futility analysis planned at 128 deaths; Test type: Superiority; p = 0.36, Log Rank; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.67 to 1.32]

2. Primary Outcome: (Phase I) Number of Subjects With Dose Limiting Toxicities (DLT) on the Two Pilot Arms
Description: Adverse events were graded using CTCAE v2.0. Grade refers to the severity of the adverse event (AE). The CTCAE v2.0 assigns Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline: Grade 1 Mild AE, Grade 2 Moderate AE, Grade 3 Severe AE, Grade 4 Life-threatening or disabling AE, Grade 5 Death related to AE. Dose limiting toxicity (DLT) was defined as grade 3+ pulmonary toxicity, grade 4+ thrombocytopenia (< 25,000 for 5 days), neutropenia (< 500/microl for 7 days), or neutropenia of any duration with fever requiring hospital admission after one dose reduction of 50% in BCNU. A 20% rate of grade 3+ pulmonary toxicities or a 40% rate of grade 4+ thrombocytopenia and neutropenia was considered unacceptable for a treatment arm combining RT, TMZ, and BCNU.
Time Frame: From start of treatment to 3 months
Population: Eligible patients who started study treatment on Pilot Arms 1 and 2
Measure: Count of Participants; unit: Participants
Arm/Group | Pilot Arm #1: RT+TMZ+BCNU | Pilot Arm #2: RT+TMZ+BCNU
Number analyzed (Participants) | 15 | 13
Participants
  Subjects with Pulmonary DLT | 1 | 0
  Subjects with Hematologic DLT | 4 | 3

3. Secondary Outcome: (Phase III) Time to Tumor Progression (TTP)
Description: Three-year rate is reported. Progression is defined as a radiographic increase in size of the lesion by > 25%, recurrence of the study lesion, or the development of new lesions, confirmed by imaging. Time to tumor progression was estimated using the cumulative incidence function (CIF) on tumor progression, with death as a competing risk. Per the protocol, the pilot arms were not included in the Phase III analyses.
Time Frame: as for outcome 1
Population: Eligible randomized patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Radiation Therapy + Temozolomide (TMZ) | RT + BCNU/CCNU
Number analyzed (Participants) | 97 | 99
months | 45.4 [35.2 to 55.0] | 54.7 [44.2 to 63.9]
Statistical Analysis 1: Comparison: Radiation Therapy + Temozolomide (TMZ) vs RT + BCNU/CCNU; Test type: Superiority; p = 0.46, Gray's test — 2-sided; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.55 to 1.16] — Reference level = RT + BCNU/CCNU

4. Secondary Outcome: (Phase III) Number of Patients With Grade 3 or Higher Toxicity
Description: Adverse events were graded using CTCAE v2.0. Grade refers to the severity of the AE. The CTCAE v2.0 assigns Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline: Grade 1 Mild AE, Grade 2 Moderate AE, Grade 3 Severe AE, Grade 4 Life-threatening or disabling AE, Grade 5 Death related to AE. The number of patients with grade or higher toxicity was calculated overall and for non-hematologic toxicity only. Per the protocol, the pilot arms were not included in the Phase III analyses.
Time Frame: as for outcome 1
Population: Eligible randomized patients who started study treatment
Measure: Number; unit: participants
Arm/Group | Radiation Therapy + Temozolomide (TMZ) | RT + BCNU/CCNU
Number analyzed (Participants) | 96 | 99
participants
  Overall toxicity | 46 | 75
  Non-hematologic toxicity | 31 | 34
Statistical Analysis 1: Comparison: Radiation Therapy + Temozolomide (TMZ) vs RT + BCNU/CCNU; Overall toxicity; Test type: Superiority; p < 0.001, Chi-squared — 2-sided
Statistical Analysis 2: Comparison: Radiation Therapy + Temozolomide (TMZ) vs RT + BCNU/CCNU; Non-hematologic toxicity; Test type: Superiority; p = 0.76, Chi-squared — 2-sided

5. Secondary Outcome: (Phase III) Survival Time by MGMT Status
Description: Survival time is defined as time from randomization to date of death from any cause and is estimated by the Kaplan-Meier method. Patients last known to be alive are censored at the date of last contact. Tumor tissue samples were analyzed for methylation status of methyl guanine methyl transferase (MGMT), classified as methylated vs. unmethylated.
Time Frame: as for outcome 1
Population: Eligible patients with MGMT data
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Methylated MGMT | Unmthylated MGMT
Number analyzed (Participants) | 36 | 22
years | 7.2 [4.5 to NA] — Not reached | 3.1 [1.5 to 8.7]
Statistical Analysis 1: Comparison: Methylated MGMT vs Unmthylated MGMT; Test type: Superiority; p = 0.08, Log Rank; Two-side significance level = 0.05; Hazard Ratio (HR) = 1.78, 95% CI 2-sided [0.93 to 3.40] — Reference level = Methylated MGMT

6. Secondary Outcome: (Phase III) Progression-free Survival by MGMT Status
Description: Progression is defined as a radiographic increase in size of the lesion by > 25%, recurrence of the study lesion, or the development of new lesions, confirmed by imaging. Progression-free survival time is defined as time from randomization to date of progression or death from any cause and is estimated by the Kaplan-Meier method. Patients last known to be alive are censored at the date of last contact. Tumor tissue samples were analyzed for methylation status of methyl guanine methyl transferase (MGMT), classified as methylated vs. unmethylated.
Time Frame: as for outcome 1
Population: Eligible patients with MGMT data
Measure: Median (95% Confidence Interval); unit: years
Groups:
- Methylated MGMT: Patients with MGMT menthylated status
Arm/Group | Methylated MGMT | Unmthylated MGMT
Number analyzed (Participants) | 36 | 22
years | 4.0 [1.4 to 7.5] | 2.1 [0.8 to 5.6]
Statistical Analysis 1: Comparison: Methylated MGMT vs Unmthylated MGMT; Test type: Superiority; p = 0.41, Log Rank; Two-sided confidence interval = 0.5; Hazard Ratio (HR) = 1.29, 95% CI 2-sided [0.70 to 2.35] — Reference level = Methylated

ADVERSE EVENTS:
Description: Eligible subjects who started study treatment and have toxicity information are included. Subjects experiencing more than one of a given adverse event are counted only once for that adverse event.
Arm/Group | Radiation Therapy + Temozolomide (TMZ) | RT + BCNU/CCNU | Pilot Arm #1: RT+TMZ+BCNU | Pilot Arm #2: RT+TMZ+BCNU
Serious Adverse Events (participants affected / at risk) | 43/96 | 72/99 | 8/15 | 11/13
Other Adverse Events (participants affected / at risk) | 94/96 | 95/99 | 14/15 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Radiation Therapy + Temozolomide (TMZ) (N=96) | RT + BCNU/CCNU (N=99) | Pilot Arm #1: RT+TMZ+BCNU (N=15) | Pilot Arm #2: RT+TMZ+BCNU (N=13)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 4 | 1 | 0
Hemoglobin decreased (Blood and lymphatic system disorders) | 1 | 14 | 3 | 0
Packed red blood cell transfusion (Blood and lymphatic system disorders) | 2 | 2 | 2 | 0
Platelet transfusion (Blood and lymphatic system disorders) | 3 | 10 | 2 | 2
Edema NOS (Cardiac disorders) | 0 | 2 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 1 | 0 | 0
Otitis externa (exc boil of meatus) NOS (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Otitis media serous NOS (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Late RT Toxicity:Eye NOS (Eye disorders) | 1 | 0 | 0 | 0
Caecitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diarrhea NOS (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 2 | 0 | 0
Vomiting NOS (Gastrointestinal disorders) | 1 | 2 | 0 | 0
Constitutional symptons-Other (General disorders) | 0 | 0 | 0 | 1
Late RT Toxicity:Other NOS (General disorders) | 0 | 0 | 0 | 1
Pain-other (General disorders) | 1 | 0 | 0 | 0
Infection NOS (Infections and infestations) | 0 | 2 | 1 | 0
Infection with grade 3 or 4 neutropenia (Infections and infestations) | 2 | 4 | 2 | 2
Infection, Other (Infections and infestations) | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 2 | 0 | 0 | 0
Bilirbin-graft versus host disease (Investigations) | 0 | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 1 | 0 | 0
Leukopenia NOS (Investigations) | 4 | 9 | 3 | 4
Lymphopenia (Investigations) | 3 | 7 | 0 | 0
Neutropenia (Investigations) | 13 | 43 | 6 | 5
Neutrophils/granulocytes for BMT (Investigations) | 1 | 0 | 0 | 0
Platelet count decreased (Investigations) | 16 | 43 | 6 | 9
Pulmonary function test NOS decreased (Investigations) | 0 | 2 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 1
Acidosis NOS (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Hyperglycemia NOS (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyperuricemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Amnesia NEC (Nervous system disorders) | 1 | 1 | 0 | 0
Ataxia NEC (Nervous system disorders) | 1 | 1 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 1 | 0 | 0
Convulsions NOS (Nervous system disorders) | 3 | 4 | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 1 | 0 | 1
Dizziness (exc vertigo) (Nervous system disorders) | 1 | 0 | 0 | 1
Headache NOS (Nervous system disorders) | 4 | 4 | 0 | 0
Hemorrhagic stroke (Nervous system disorders) | 2 | 0 | 0 | 0
Late RT Toxicity:Brain NOS (Nervous system disorders) | 1 | 1 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 6 | 2 | 0 | 1
Speech disorder NEC (Nervous system disorders) | 1 | 2 | 0 | 0
Syncope (Nervous system disorders) | 2 | 0 | 0 | 0
Vertigo NEC (Nervous system disorders) | 0 | 0 | 1 | 0
Depression NEC (Psychiatric disorders) | 0 | 1 | 0 | 0
Euphoric mood (Psychiatric disorders) | 1 | 0 | 0 | 0
Personality change (Psychiatric disorders) | 1 | 0 | 0 | 0
Renal failure NOS (Renal and urinary disorders) | 0 | 1 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0 | 0
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dyspnea NOS (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary-other (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Culture wound positive (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Dermatitis exfoliative NOS (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Hypertension NOS (Vascular disorders) | 1 | 0 | 0 | 0
Thrombosis NOS (Vascular disorders) | 2 | 2 | 1 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Radiation Therapy + Temozolomide (TMZ) (N=96) | RT + BCNU/CCNU (N=99) | Pilot Arm #1: RT+TMZ+BCNU (N=15) | Pilot Arm #2: RT+TMZ+BCNU (N=13)
Hematologic-Other (Blood and lymphatic system disorders) | 4 | 5 | 0 | 1
Hemoglobin decreased (Blood and lymphatic system disorders) | 32 | 59 | 13 | 13
Edema NOS (Cardiac disorders) | 3 | 6 | 0 | 2
Hearing impaired (Ear and labyrinth disorders) | 5 | 9 | 0 | 1
Hearing-Other (Ear and labyrinth disorders) | 8 | 6 | 0 | 1
Vision blurred (Eye disorders) | 12 | 10 | 2 | 1
Constipation (Gastrointestinal disorders) | 37 | 8 | 3 | 0
Diarrhea NOS (Gastrointestinal disorders) | 13 | 12 | 1 | 1
Dry mouth (Gastrointestinal disorders) | 5 | 5 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 9 | 5 | 0 | 1
Esophagitis NOS (Gastrointestinal disorders) | 5 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 75 | 42 | 7 | 7
Stomatitis (Gastrointestinal disorders) | 9 | 3 | 1 | 0
Vomiting NOS (Gastrointestinal disorders) | 34 | 16 | 3 | 1
Fatigue (General disorders) | 78 | 73 | 9 | 9
Late RT Toxicity:Other NOS (General disorders) | 17 | 17 | 4 | 3
Pain-other (General disorders) | 9 | 11 | 0 | 2
Pyrexia (General disorders) | 2 | 6 | 0 | 0
Infection NOS (Infections and infestations) | 10 | 6 | 0 | 0
Late RT Toxicity:Skin(within RT field)NOS (Injury, poisoning and procedural complications) | 13 | 11 | 3 | 1
Alanine aminotransferase increased (Investigations) | 22 | 21 | 3 | 2
Aspartate aminotransferase increased (Investigations) | 21 | 18 | 5 | 1
Blood alkaline phosphatase NOS increased (Investigations) | 13 | 18 | 2 | 2
Leukopenia NOS (Investigations) | 37 | 70 | 12 | 10
Lymphopenia (Investigations) | 15 | 13 | 0 | 0
Metabolic-Other (Investigations) | 5 | 4 | 0 | 1
Neutropenia (Investigations) | 17 | 45 | 4 | 2
Platelet count decreased (Investigations) | 44 | 63 | 9 | 11
Pulmonary function test NOS decreased (Investigations) | 0 | 9 | 5 | 3
Weight decreased (Investigations) | 10 | 10 | 2 | 3
Anorexia (Metabolism and nutrition disorders) | 31 | 23 | 6 | 3
Hyperglycemia NOS (Metabolism and nutrition disorders) | 9 | 7 | 1 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 7 | 7 | 4 | 2
Hypokalemia (Metabolism and nutrition disorders) | 6 | 5 | 3 | 2
Hyponatremia (Metabolism and nutrition disorders) | 3 | 6 | 4 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 2 | 1 | 1
Muscle weakness NOS (Musculoskeletal and connective tissue disorders) | 12 | 5 | 1 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 4 | 0 | 0
Amnesia NEC (Nervous system disorders) | 14 | 13 | 2 | 2
Ataxia NEC (Nervous system disorders) | 4 | 5 | 0 | 2
Convulsions NOS (Nervous system disorders) | 13 | 13 | 2 | 3
Dizziness (exc vertigo) (Nervous system disorders) | 16 | 13 | 0 | 2
Headache NOS (Nervous system disorders) | 45 | 31 | 2 | 7
Late RT Toxicity:Brain NOS (Nervous system disorders) | 11 | 14 | 3 | 4
Learning disorder NOS (Nervous system disorders) | 5 | 3 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 11 | 7 | 1 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 14 | 9 | 1 | 1
Speech disorder NEC (Nervous system disorders) | 8 | 4 | 0 | 0
Taste disturbance (Nervous system disorders) | 14 | 13 | 3 | 1
Tremor NEC (Nervous system disorders) | 7 | 4 | 1 | 2
Anxiety NEC (Psychiatric disorders) | 12 | 9 | 1 | 1
Confusion (Psychiatric disorders) | 2 | 10 | 2 | 1
Depression NEC (Psychiatric disorders) | 12 | 6 | 1 | 2
Insomnia NEC (Psychiatric disorders) | 18 | 8 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 7 | 0 | 1
Dyspnea NOS (Respiratory, thoracic and mediastinal disorders) | 7 | 13 | 0 | 5
Alopecia (Skin and subcutaneous tissue disorders) | 56 | 58 | 6 | 9
Dermatitis exfoliative NOS (Skin and subcutaneous tissue disorders) | 13 | 7 | 2 | 0
Dermatitis radiation NOS (Skin and subcutaneous tissue disorders) | 17 | 16 | 2 | 1
Injection site reaction NOS (Skin and subcutaneous tissue disorders) | 0 | 8 | 0 | 2
Skin-Other (Skin and subcutaneous tissue disorders) | 6 | 2 | 0 | 0
Phlebitis superficial (Vascular disorders) | 0 | 5 | 0 | 0

LIMITATIONS AND CAVEATS:
Accrual to the TMZ BCNU arm required an acceptable toxicity profile from a pilot arm. Treatment cessation/reduction for toxicity caused the combination arm to be dropped. Per the protocol, the pilot arms were not included in the Phase III analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI's are required to abide by the sponsor's publication guidelines which require review by coauthors and subsequent review and approval by the sponsor.